CLINICAL TRIAL: NCT06939114
Title: Optic Nerve Sonography to Monitor Intracranial Pressure After Ischemic sTrokE - The ONSITE Study
Acronym: ONSITE
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Susanne Wegener, Prof. Dr. med., University of Zurich
Other Study IDs: 2018-01946
Record Dates: First submitted 2025-04-04; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Malignant Media Infarction; Stroke; Intracranial Hypertension
Keywords: Stroke; Ischemic Stroke; Ultrasound; Optic nerve sheath; Optic nerve sheath diameter; Malignant media infarction; Intracranial pressure; Intracranial hypertension; Large vessel occlusion stroke
MeSH Terms: conditions — Stroke; Intracranial Hypertension; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stroke: Patient with acute ischemic stroke
- Non-Stroke, non-IH controls: Patient without acute stroke or history of intracranial hypertension

SUMMARY:
The goal of the ONSITE study is to investigate whether an increase Optic nerve sheath diameter (ONSD) may help to predict intracranial hypertension (IH) after stroke. IH is a life-threatening complicaitons of malignant middle cerebral artery (MCA) infarction due to space-occupying brain edema. Patients at risk are monitored based on clinical symptoms, which can be difficult due to comorbidities such as delirium or systemic infections, which can hempen clinical judgement. Readily available, non-invasive methods to monitor ICP in stroke patients could help to earlier diagnose rising ICP and facilitate treatment decisions such as hemicraniectomy. This study investigates whether ONSD with optic nerve sonography (ONS) can detect brain edema after stroke.

DETAILED DESCRIPTION:
Intracranial Hypertension (IH) is a life-threatening complication after ischemic and hemorrhagic stroke. IH develops in ischemic stroke due to brain edema, which may occur in large-vessel occlusion, most common in large middle cerebral artery (MCA) infarcts due to occlusion of the internal carotid artery (ICA) or occlusion of the proximal segment (M1) of the middle cerebral artery. Up to 30% of patients with occlusion of these vessels develop large space-occupying brain edema leading to a serious condition termed "malignant media infarction" leading to rapid neurological deterioration and reduced consciousness. IH usually develops within the first 24-96 hours after stroke; however, the exact time course is not predictable.

IH is a life-threatening emergency that demands immediate medical or surgical action. As it is not possible to predict the course of intracerebral pressure increase in patients at risk, it is necessary to monitor these patients closely. However, clinical observation of neurological symptoms may be hampered, as stroke patients often require pain or anxiolytic medications or suffer from typical comorbidities of stroke, such as infection, cardiac diseases, or delirium, which limit judgment of neurological symptoms. Despite the limitations of clinical symptom prediction for IH, ICP is not routinely monitored in stroke patients as invasive intracranial devices, the current gold standard for ICP monitoring have several drawbacks that limit their routine application. Intracranial ICP monitors require a neurosurgical intervention, which may not always be feasible or contraindicated in several conditions such as coagulopathy and thrombocytopenia. Furthermore, ICP monitors are associated with complications such as hemorrhages (1.1-5.8% of cases), infection (0-15% of cases) or monitor malfunction (6.3-40% of cases).

Because of these limitations, noninvasive methods to measure ICP have been eagerly sought. Se-rial computer tomography (CT) or Magnetic Resonance Imaging (MRI) are applied to detect in-creased ICP in patients at risk. However, imaging is expensive, potential harmful to patients due to radiation or necessity to lie supine and still for a prolonged period and have limited availability. As such, their use is restricted as well. Furthermore there are studies suggesting that CT scans might have a poor sensitivity for detection of IH.

Ultrasonography is an alternative tool to measure ICP non-invasively. Ultrasonography is a low cost, simple bedside tool, widely available in emergency rooms as well as on stroke units. Optic nerve sonography (ONS) to measure the optic nerve sheath diameter (ONSD) has been developed and suggested as an alternative sonographic method to detect IH. ONS utilizes the fact that the optic nerve sheath, which is readily visualized by transorbital ultrasound, is filled with spinal fluid and grows in diameter according to ICP. To perform ONS, the patient is placed in a position 20̊ supine to horizontal. The probe is then placed on the temporal side of the closed eyelid without pressure to avoid any damage to the eye. The position of the probe is then adjusted until the entry of the optic nerve into the globe of the eye is visible. ONSD is measured 3 mm behind the globe, as this position shows the greatest distension of the optic sheath in IH patients and thus has become the standard measurement point.

The method is quickly learned and a trained operator can perform measurement of ONSD in both eyes in less than 4 minutes. In current clinical practice, ONS has been used in intensive care setting to monitor ICP and diagnose brain death in brain trauma patients. ONS is also used in other neurological diseases, such as idiopathic intracranial hypertension. It was shown in several studies, as well as meta-analyses that ONS derived measurements of intracranial hypertension can be performed with good intra- and interobserver reliability. In a meta-analysis, in which ONDS was compared to invasive ICP measurements, ONSD showed good test accuracy with a pooled sensitivity of 90% and pooled specificity of 85%. When compared to CT scan, ONSD showed good accuracy for IH as well, with a sensitivity of 95.6% and specificity of 92.3%. ONSD can also be used to rapidly assess the success of therapeutic interventions. For example, patients with idiopathic intracranial hypertension showed a significantly reduced ONSD directly af-ter lumbar puncture with therapeutic removal of 30-50 ml of cerebrospinal fluid (CSF).

Several studies raised the question of which cut-off value should be used for the ONSD in healthy individuals. Earlier studies that compared ONSD to CT results suggested a upper normal value of 4.5 mm for individuals aged ≤1 year and 5.0 mm for those aged >1 year. More recent studies, however, comparing ONSD to invasive ICP measurements, suggested that a cut-off value of 5.7-6.0mm provided the best accuracy and that values above that cut off should alert the clinician of IH.

Preliminary data from routine evaluation of ONSD in patients with stroke and ICH showed significantly increased ONSD on the side of stroke compared to the contralateral side. The investigators also tested for the feasibility of the method in patients with diagnosed idiopathic intracranial hyper-tension, which were found to have larger ONSD than healthy individuals on both sides. In each patient, 3 individual measurements per eye were averaged.

The goal of this study is to improve stroke patient care by helping to investigate whether ONS is a feasible tool to diagnose IH after stroke, as IH is one of the most troublesome and life-threatening complications of large-vessel ischemic stroke. It is critical that the clinician does not miss rising ICP so that life-saving treatment is not delayed. ONS measurement of ICP is an accurate, widely avail-able and easy to learn method to detect IH and has been successfully used in clinical practice in several fields of neurology. Its value in acute stroke care, however, remains uncertain. The investigators have tested ONS derived ONSD measurements and have confirmed the feasibility to use this parameter. If ONSD thresholds can be established to detect IH early after stroke, it could be further tested in a clinical trial to aid in decision making for hemicraniectomy in stroke patients.

This study aims to investigate the hypothesis that ONS is a feasible method to detect IH in stroke patients. To this end, the primary objective is to observe the changes in ONSD after large-vessel ischemic stroke and in the presence of IH.

The second objective is to derive a cut-off value for ONSD that best predicts the presence of IH in stroke patients and to assess whether this cut-off value would be able to detect IH before clinical changes occur (assessed by the Glasgow Coma Scale (GCS) and/or National Institutes of Health Stroke Scale (NIHSS) in patients at risk). This cut-off value could be the base for a future clinical trial to evaluate the diagnostic performance of this method in stroke patients. In addition, the investigators aim to investigate the predictive value of the ONSD in the clinical outcome after stroke (as derived from the modified Rankin Scale (mRS) and NIHSS after 3 month).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Consent according to the regulations of research in an emergency situation
* For non-Control patients: Acute ischemic stroke within 24 hours of recruitment

Exclusion Criteria:

* Known intracranial space-occupying lesion
* Known history of intracranial hypertension
* Contra-indications on ethical grounds
* Expected or known non-compliance to participate in the observational study, severe drug- or/and alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For non-stroke, non-IH patients we will recruit patients hospitalized at the Department of Neurology, University Hospital of Zurich. Patients within the clinic are screened for inclusion / exclusion criteria. If a patient is considered eligible for the study, he or she will be contacted by a member of the study team.
  For stroke patients acute stroke patients admitted to the Department of Neurology, University Hospital of Zurich will be screened for study eligibility. If a patient is considered eligible for the study, he or she will be contacted by a member of the study team after initial emergency care is completed.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Presence of intracranial hypertension | Assessed at Baseline, at 12 hours after stroke, at 24 hours after stroke, at 36 hours after stroke, at 48 hours after stroke, at 72 hours after stroke, at 120 hours after stroke.
  Intracranial hypertension is defined in our study as midline shift ≥ 3mm or a decrease in GCS without any other cause based on clinical judgement or patient requiring hemicraniectomy.

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | Obtained at Baseline, at 12 hours after stroke, at 24 hours after stroke, at 36 hours after stroke, at 48 hours after stroke, at 72 hours after stroke, at 120 hours after stroke, at 3 months after stroke
  The National Institutes of Health Stroke Scale (NIHSS) is a 11-point neurological exam used to quantify the severity of an acute stroke. The NIHSS assesses level of consciousness, eye move-ments, visual fields, facial muscle function, extremity strength, sensory function, coordination, language, speech, and neglect. It is a commonly used tool in clinical routine, as well as in stroke re-search.
Glasgow Coma Scale (GCS) | Obtained at Baseline, at 12 hours after stroke, at 24 hours after stroke, at 36 hours after stroke, at 48 hours after stroke, at 72 hours after stroke, at 120 hours after stroke, at 3 months after stroke
  The Glasgow Coma Scale (GCS) is a 3-point neurological exam used to assess the level of con-sciousness of a patient. The GCS consists of an assessment of eye response, verbal response and motor response.
modified Rankin Scale (mRS) | mRS is measured 3 months after stroke
  The modified Rankin Scale (mRS) is a widely used scale of measuring the degree of disability of people who have suffered a stroke. The mRS is used in clinical practice, as well as in stroke studies to describe the clinical outcome after stroke. The mRS runs from 0 to 6, with 0 being a patient with-out any disability and 6 indicating for death of the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Will be decided upon reasonable request

REFERENCES:
- [Background] Bauerle J, Nedelmann M. Sonographic assessment of the optic nerve sheath in idiopathic intracranial hypertension. J Neurol. 2011 Nov;258(11):2014-9. doi: 10.1007/s00415-011-6059-0. Epub 2011 Apr 28. PMID 21523461
- [Background] Bauerle J, Lochner P, Kaps M, Nedelmann M. Intra- and interobsever reliability of sonographic assessment of the optic nerve sheath diameter in healthy adults. J Neuroimaging. 2012 Jan;22(1):42-5. doi: 10.1111/j.1552-6569.2010.00546.x. Epub 2010 Dec 1. PMID 21121998
- [Background] Toscano M, Spadetta G, Pulitano P, Rocco M, Di Piero V, Mecarelli O, Vicenzini E. Optic Nerve Sheath Diameter Ultrasound Evaluation in Intensive Care Unit: Possible Role and Clinical Aspects in Neurological Critical Patients' Daily Monitoring. Biomed Res Int. 2017;2017:1621428. doi: 10.1155/2017/1621428. Epub 2017 Mar 21. PMID 28421189
- [Background] Tayal VS, Neulander M, Norton HJ, Foster T, Saunders T, Blaivas M. Emergency department sonographic measurement of optic nerve sheath diameter to detect findings of increased intracranial pressure in adult head injury patients. Ann Emerg Med. 2007 Apr;49(4):508-14. doi: 10.1016/j.annemergmed.2006.06.040. Epub 2006 Sep 25. PMID 16997419
- [Background] Ohle R, McIsaac SM, Woo MY, Perry JJ. Sonography of the Optic Nerve Sheath Diameter for Detection of Raised Intracranial Pressure Compared to Computed Tomography: A Systematic Review and Meta-analysis. J Ultrasound Med. 2015 Jul;34(7):1285-94. doi: 10.7863/ultra.34.7.1285. PMID 26112632
- [Background] Hansen HC, Helmke K. The subarachnoid space surrounding the optic nerves. An ultrasound study of the optic nerve sheath. Surg Radiol Anat. 1996;18(4):323-8. doi: 10.1007/BF01627611. PMID 8983112
- [Background] Hansen HC, Helmke K. Validation of the optic nerve sheath response to changing cerebrospinal fluid pressure: ultrasound findings during intrathecal infusion tests. J Neurosurg. 1997 Jul;87(1):34-40. doi: 10.3171/jns.1997.87.1.0034. PMID 9202262
- [Background] Galetta S, Byrne SF, Smith JL. Echographic correlation of optic nerve sheath size and cerebrospinal fluid pressure. J Clin Neuroophthalmol. 1989 Jun;9(2):79-82. PMID 2526162
- [Background] Dubourg J, Javouhey E, Geeraerts T, Messerer M, Kassai B. Ultrasonography of optic nerve sheath diameter for detection of raised intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2011 Jul;37(7):1059-68. doi: 10.1007/s00134-011-2224-2. Epub 2011 Apr 20. PMID 21505900
- [Background] Ropper AH, Shafran B. Brain edema after stroke. Clinical syndrome and intracranial pressure. Arch Neurol. 1984 Jan;41(1):26-9. doi: 10.1001/archneur.1984.04050130032017. PMID 6606414
- [Background] Schwab S, Aschoff A, Spranger M, Albert F, Hacke W. The value of intracranial pressure monitoring in acute hemispheric stroke. Neurology. 1996 Aug;47(2):393-8. doi: 10.1212/wnl.47.2.393. PMID 8757010
- [Background] Wijdicks EF, Sheth KN, Carter BS, Greer DM, Kasner SE, Kimberly WT, Schwab S, Smith EE, Tamargo RJ, Wintermark M; American Heart Association Stroke Council. Recommendations for the management of cerebral and cerebellar infarction with swelling: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Apr;45(4):1222-38. doi: 10.1161/01.str.0000441965.15164.d6. Epub 2014 Jan 30. PMID 24481970
- [Background] Heiss WD. Malignant MCA Infarction: Pathophysiology and Imaging for Early Diagnosis and Management Decisions. Cerebrovasc Dis. 2016;41(1-2):1-7. doi: 10.1159/000441627. Epub 2015 Nov 19. PMID 26581023
- [Background] Hacke W, Schwab S, Horn M, Spranger M, De Georgia M, von Kummer R. 'Malignant' middle cerebral artery territory infarction: clinical course and prognostic signs. Arch Neurol. 1996 Apr;53(4):309-15. doi: 10.1001/archneur.1996.00550040037012. PMID 8929152
- [Background] Hofmeijer J, Algra A, Kappelle LJ, van der Worp HB. Predictors of life-threatening brain edema in middle cerebral artery infarction. Cerebrovasc Dis. 2008;25(1-2):176-84. doi: 10.1159/000113736. Epub 2008 Jan 23. PMID 18212524